CLINICAL TRIAL: NCT05470972
Title: Endometrioma Cystic Fluid Aspiration and Retained Ethanol Sclerotherapy Might Improve the Systemic Immune Milieu
Brief Title: Relation Between Ethanol Sclerotherapy for Endometrioma Systemic Immune Milieu
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Hagars, Assistant professor of gynecology, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35560/6/22
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian Endometrioma (Experimental): Ovarian endometrioma (OE) is in women of reproductive age
  Interventions: Drug: Ethanol Injection

INTERVENTIONS:
Drug: Ethanol Injection — The AEST procedure was performed as follows: vaginal walls were cleansed using vaginal povidone-iodine, a 17 gauge, 30-cm length needle was inserted through the posterior vaginal fornix into the pouch of Douglas, and the cyst was aspirated till complete disappearance of the cyst on the ultrasound scanner. The collected cystic fluid was collected into a plastic tube without an anticoagulant. The needle was maintained in its place, the syringe was removed and the cyst was flushed with saline solution until obtaining a clear liquid. Then, 96% ethanol was injected as 60% of the volume of the aspirated fluid to guard against over distension or rupture of the cyst and/or ethanol diffusion into the pelvis. The collected fluid was divided into three sterile tubes for cytological and bacteriological examinations and the study investigations. Patients were allowed to be completely recovered and were discharged home.

SUMMARY:
Design: Prospective interventional study. 69 women with OE were evaluated clinically and by transvaginal ultrasonography (TUV). AEST procedure was performed and the collected aspirate and pre-procedural blood samples were collected for estimation of cytokines' levels. At 6-m post-procedure, clinical evaluation and TUV were repeated and serum cytokines' levels were re-estimated.

ELIGIBILITY:
Inclusion Criteria:

* Women with OE of a mean diameter of >3 cm

Exclusion Criteria:

* Women with recurrent OE
* a cyst that was suspicious of being malignant
* diabetes mellitus
* polycystic ovary syndrome
* body mass index (BMI) of >30 kg/m2
* previous surgical interference that resulted in pelvic adhesions

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
The effect of AEST procedures on patients' cytokines levels. | 6 months
  The effect of AEST on patients serum levels of tumor necrosis factor-α, interleukin-8 and interleukin-10

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, El-Gharbyia, Egypt